CLINICAL TRIAL: NCT04001894
Title: Ticagrelor and Clopidogrel on Platelet Effects in Chinese Patients With Stable Coronary Artery Disease: a Randomized, Single-blind, Crossover Clinical Study
Brief Title: Ticagrelor and Clopidogrel on Platelet Effects in Chinese Patients With Stable Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yue LI, Professor, First Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20190515
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Platelet Reactivity
Keywords: Ticagrelor; Clopidogrel; Coronary artery disease; platelet function tests
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor (Experimental): To observe the safety and efficacy of standard-dose ticagrelor in Chinese patients with Stable Coronary Artery Disease
  Interventions: Drug: Ticagrelor 90mg; Drug: Clopidogrel 75mg
- Clopidogrel (Active Comparator): To observe the safety and efficacy of standard-dose clopidogrel in Chinese patients with Stable Coronary Artery Disease
  Interventions: Drug: Ticagrelor 90mg; Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Ticagrelor (90.0 mg twice daily) for 2 weeks, followed by a 2-week washout period then 2 weeks crossover phase of clopidogrel (75mg once daily).
  Other Names: Ticagrelor
Drug: Clopidogrel 75mg — Clopidogrel (75mg once daily) for 2 weeks, followed by a 2-week washout period then 2 weeks crossover phase of ticagrelor (90.0 mg twice daily).
  Other Names: Clopidogrel

SUMMARY:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 inhibitor reduces thrombotic events in patients with coronary artery disease, but these benefits come at the expense of increased risk of bleeding when compared with aspirin monotherapy. Increased evidence showed that P2Y12 inhibitor monotherapy still maintain antiischemic efficacy while reducing the bleeding risk compared with DAPT. Therefore, the investigators performed this study to observe the efficacy of ticagrelor in comparison to clopidogrel in Chinese patients with stable CAD.

DETAILED DESCRIPTION:
Ticagrelor is a novel, direct-acting, reversibly binding P2Y12 receptor antagonist. When related with clopidogrel, ticagrelor exhibits a more potent and more predictable antiplatelet effect with a faster onset and offset of action. Current guidelines give a recommendation on the use of dual antiplatelet therapy support ticagrelor 90 mg twice daily over clopidogrel 75 mg daily in addition to aspirin in CAD patients. However, increasing evidence showed ticagrelor increased the risk of bleeding. Recent studies showed that P2Y12 inhibitor monotherapy still maintain antiischemic efficacy while reducing the bleeding risk compared with DAPT. So the investigators performed this randomized, single-blind, crossover clinical trial to observe the effects of standard-dose ticagrelor and standard-dose clopidogrel on platelet reactivity in Chinese patients with stable CAD.

ELIGIBILITY:
Inclusion Criteria:•

* Aged ≥18 years
* Subjects had documented with stable CAD
* Women were required to be postmenopausal or surgically sterile
* Patients were required to discontinue clopidogrel or ticagrelor at least 14 days before randomization
* Patients were required to discontinue aspirin at least 14 days before randomization.

Exclusion Criteria:

* Acute coronary syndrome
* Planned use of glycoprotein IIb/IIIa receptor inhibitors, adenosine diphosphate (ADP) receptor antagonists other than the study medication, or anticoagulant therapy during the study period
* Platelet count <10×10^4/μL
* Hstory of bleeding tendency
* Diagnosed as respiratory or circulatory instability
* Allergy to ticagrelor or clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
The platelet inhibition ratio | up to 3 months
  Thromboelastogram was used to measure platelet inhibition ratio.

SECONDARY OUTCOMES:
The platelet aggregation ratio. | up to 3 months
  Light transmittance aggregometry method was used to measure platelet aggregation ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Li, Doctor, Principal Investigator — First Affiliated Hospital of Harbin Medical University
Locations (1):
- Thrombelastogram, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No